CLINICAL TRIAL: NCT00465985
Title: A Three-part,Multicenter Study,With a Randomized,Double-blind,Placebo Controlled,Withdrawal Design in Part II to Assess Efficacy,Safety,and Tolerability of ACZ885(Anti-interleukin-1beta Monoclonal Antibody)in Patients With Muckle-Wells Syndrome
Brief Title: Efficacy, Safety, and Tolerability of ACZ885 in Patients With Muckle-Wells Syndrome
Acronym: REMITTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CACZ885D2304
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2011-02-11 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Muckle Wells Syndrome
Keywords: Muckle-Wells Syndrome; children; systemic autoinflammatory disease; CIAS-1 gene; NALP-3; ACZ885; human monoclonal anti-human interleukin-1beta (IL-1beta); antibody; autosomal dominant; familial autoinflammatory syndrome
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Part I, Part II-arm1, & Part III (Experimental)
  Interventions: Drug: ACZ885
- Part II - arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACZ885
  Arms: Part I, Part II-arm1, & Part III
Drug: Placebo
  Arms: Part II - arm 2

SUMMARY:
This study is designed to provide efficacy and safety data for ACZ885 (a fully human anti-interleukin-1beta (anti-IL-1beta) monoclonal antibody) administered as an injection subcutaneously (s.c.) in patients with Muckle-Wells Syndrome.

Part I is an 8-week open-label, active treatment period to identify ACZ885 responders.

Part II is a double-blind, placebo-controlled period to assess primarily the efficacy of ACZ885 compared to placebo.

Part III is an open-label, active treatment period where patients will receive ACZ885 every 8 weeks after withdrawal or completion of Part II.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of NALP3 mutations and clinical picture resembling Muckle-Wells Syndrome.
* Muckle-Wells Syndrome patients who participated in the CACZ885A2102 study, will have the option to participate in this study upon disease flare
* Muckle-Wells Syndrome patients requiring medical intervention either untreated or treated (i.e. under ACZ885, anakinra, or any other investigational IL-1 blocking therapy).

Exclusion Criteria:

* History of being immunocompromised, including a positive HIV at screening test result.
* No live vaccinations within 3 months prior to the start of the trial, during the trial, and up to 3 months following the last dose.
* History of significant medical conditions, which in the Investigator's opinion would exclude the patient from participating in this trial.
* History of recurrent and/or evidence of active bacterial, fungal, or viral infections.
* Positive tuberculin skin test at 48 to 72 hours after administration at the screening visit or within 2 months prior to the screening visit, according to national guidelines.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (3):
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Madison, Wisconsin
- France (5):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigational Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Tübingen, Germany
- Novartis Investigative Site, New Delhi, India
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, London, United Kingdom

REFERENCES:
- [Derived] Kone-Paut I, Lachmann HJ, Kuemmerle-Deschner JB, Hachulla E, Leslie KS, Mouy R, Ferreira A, Lheritier K, Patel N, Preiss R, Hawkins PN; Canakinumab in CAPS Study Group. Sustained remission of symptoms and improved health-related quality of life in patients with cryopyrin-associated periodic syndrome treated with canakinumab: results of a double-blind placebo-controlled randomized withdrawal study. Arthritis Res Ther. 2011;13(6):R202. doi: 10.1186/ar3535. Epub 2011 Dec 9. PMID 22152723
- [Derived] Lachmann HJ, Kone-Paut I, Kuemmerle-Deschner JB, Leslie KS, Hachulla E, Quartier P, Gitton X, Widmer A, Patel N, Hawkins PN; Canakinumab in CAPS Study Group. Use of canakinumab in the cryopyrin-associated periodic syndrome. N Engl J Med. 2009 Jun 4;360(23):2416-25. doi: 10.1056/NEJMoa0810787. PMID 19494217

RESULTS

PARTICIPANT FLOW:
Groups:
- ACZ885: ACZ885 150 mg subcutaneous injection or 2 mg/kg subcutaneous injection, depending on body weight, every 8 weeks.
- Placebo: Placebo subcutaneous injection every 8 weeks.
Period: Part I - Open-label Treatment Period
Arm/Group | ACZ885 | Placebo
Started | 35 (All patients received treatment with ACZ885 in Part I of the study.) | 0
Completed | 31 (Only patients with a complete response completed Part I and entered Part II of the study.) | 0
Not Completed | 4 | 0
Not completed — Unsatisfactory therapeutic effect | 4 | 0
Period: Part II - 1:1 ACZ885:Placebo
Arm/Group | ACZ885 | Placebo
Started | 15 (Patients with complete response to treatment entered Part II and were randomized to ACZ885 ,placebo.) | 16
Completed | 15 | 4
Not Completed | 0 | 12
Not completed — Unsatisfactory therapeutic effect | 0 | 12
Period: Part III - Open-label Treatment Period
Arm/Group | ACZ885 | Placebo
Started | 31 (All patients received treatment with ACZ885 in Part III of the study.) | 0
Completed | 29 | 0
Not Completed | 2 | 0
Not completed — Unsatisfactory therapeutic effect | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | ACZ885
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Disease Flare in Part II (After 24 Weeks of the Double-blind Part)
Description: Determined by the Physician's global assessment of autoinflammatory disease activity, assessment of skin disease and inflammation markers. Data expressed as a percent of participants who had experienced a flare by the end of Part II.
Time Frame: 32 weeks after study start
Measure: Number; unit: percent of participants
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 15 | 16
percent of participants | 0 | 81.3

2. Secondary Outcome: Number of Participants With Treatment Response in Part I (After 8 Weeks)
Description: Treatment response was based on Physician's global assessment(PGA) of autoinflammatory disease activity, assessment of skin disease(SD) and serum values of C-reactive protein(CRP) and/or serum amyloid A(SAA). Complete Response (CR):PGA and SD ≤ minimal and normal CRP and/or SAA. Partial Response (PR): a reduction of CRP and/or SAA from baseline (BL) by >30% but not reaching normal values and PGA improvement from BL by at least one category. Disease flare: a CRP and/or SAA > 30 mg/L and either PGA > minimal or PGA = minimal and SD > minimal. Non-responders = no PR by Day 8 or no CR by Day 15.
Time Frame: 8 weeks after study start
Measure: Number; unit: Participants
Arm/Group | ACZ885
Number analyzed (Participants) | 35
Participants
  Complete response | 31 (25.200)
  Partial response | 2
  Disease flare | 1
  Non-responder (protocol violation) | 1

3. Secondary Outcome: Investigator's Clinical Assessment of Autoinflammatory Disease Activity & Participant's Assessment of Symptoms at End of Part II (After 24 Weeks of the Double-blind Part)
Description: A 5-point scale was used for the Physician's global assessment on autoinflammatory disease activity (absent, minimal, mild, moderate and severe) and for the assessment of the following items:
  * skin disease (urticarial skin rash)
  * arthralgia
  * myalgia
  * headache/migraine
  * conjunctivitis
  * fatigue/malaise
  * other symptoms related to autoinflammatory syndrome
  * other symptoms not related to autoinflammatory syndrome
Time Frame: 32 weeks after study start
Measure: Number; unit: Participants
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 15 | 16
Participants
  Absent | 8 | 0
  Minimal | 7 | 4
  Mild | 0 | 8
  Moderate | 0 | 4
  Severe | 0 | 0

4. Secondary Outcome: Change in Inflammation Markers at the End of Part II (C-reactive Protein and/or Serum Amyloid A) (After 24 Weeks of the Double-blind Part) From Week 8.
Time Frame: Week 8 and Week 32
Population: Intention to treat (ITT)population and LOCF.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 15 | 16
mg/L
  C reactive protein (CRP (mg/L)) | 1.10 (3.086) | 19.93 (24.175)
  Serum amyloid A (SAA (mg/L)) | 2.27 (8.604) | 71.09 (136.637)

5. Secondary Outcome: Pharmacokinetics (CLD (L/d))
Description: Assessed serum clearance of ACZ885.
Time Frame: 48 weeks after study start
Population: Patients in Part I and Part II who received at least one dose of ACZ885.
Measure: Mean (Standard Deviation); unit: L/day
Arm/Group | ACZ885
Number analyzed (Participants) | 35
L/day | 0.177 (0.085)

6. Primary Outcome: Number of Participants Who Experienced a Disease Flare in Part II
Description: Disease flare is determined by the Physician's global assessment of autoinflammatory disease activity, assessment of skin disease and inflammation markers. Disease Flare = the C-reactive protein and/or serum amyloid A (SAA) > 30 mg/L and either a PGA > minimal, or PGA equal to minimal and > minimal SD.
Time Frame: 32 weeks after study start
Measure: Number; unit: Participants
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 15 | 16
Participants | 0 | 13

7. Secondary Outcome: Pharmacodynamics Measured by Interleukin-1β (IL-1β) Concentrations at End of Part I.
Time Frame: until Week 8
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ACZ885
Number analyzed (Participants) | 35
pg/mL | 19.047 (17.6609)

8. Secondary Outcome: Pharmacodynamics Measured by Interleukin-1β (IL-1β) Concentrations at End of Part II.
Time Frame: 32 weeks after study start
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ACZ885 | Placebo
Number analyzed (Participants) | 15 | 16
pg/mL | 21.943 (10.3698) | 0.596 (0.7289)

9. Secondary Outcome: Pharmacodynamics Measured by Interleukin-1β (IL-1β) Concentrations at End of Part III.
Time Frame: 48 weeks after study start
Population: Intention to treat (ITT) population.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ACZ885
Number analyzed (Participants) | 31
pg/mL | 23.018 (16.5193)

ADVERSE EVENTS:
Time Frame: 48 weeks
Groups:
- Part I ACZ885; Part II ACZ885; Part III ACZ885: ACZ885 150 mg subcutaneous injection or 2 mg/kg subcutaneous injection, depending on body weight, every 8 weeks.
- Part II Placebo: Placebo subcutaneous injection every 8 weeks.
- Entire Study ACZ885: Entire study ACZ885. The SAE and AEs were collected and reported for all three periods.
Arm/Group | Part I ACZ885 | Part II ACZ885 | Part II Placebo | Part III ACZ885 | Entire Study ACZ885
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/15 | 0/16 | 2/31 | 2/35
Other Adverse Events (participants affected / at risk) | 27/35 | 15/15 | 14/16 | 24/31 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part I ACZ885 (N=35) | Part II ACZ885 (N=15) | Part II Placebo (N=16) | Part III ACZ885 (N=31) | Entire Study ACZ885 (N=35)
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Intraocular pressure increased (Investigations) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I ACZ885 (N=35) | Part II ACZ885 (N=15) | Part II Placebo (N=16) | Part III ACZ885 (N=31) | Entire Study ACZ885 (N=35)
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 2 | 3
Erythema of eyelid (Eye disorders) | 0 | 1 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 5 | 7
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 5
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Asthenia (General disorders) | 2 | 1 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
Hangover (General disorders) | 0 | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0 | 1
House dust allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 0 | 4
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 2 | 4
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 1 | 2 | 3 | 0 | 6
Nasopharyngitis (Infections and infestations) | 4 | 4 | 2 | 4 | 12
Oral herpes (Infections and infestations) | 1 | 0 | 2 | 0 | 3
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 2 | 4
Rhinitis (Infections and infestations) | 4 | 1 | 2 | 0 | 6
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1 | 2
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 3
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 1
Weight increased (Investigations) | 3 | 0 | 0 | 1 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Complex regional pain syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 3 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 1 | 0 | 2 | 2
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2
Stress (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 3
Haematoma (Vascular disorders) | 1 | 0 | 1 | 0 | 2
Hot flush (Vascular disorders) | 1 | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The outcomes for this study were reported in separate tables for each period. The SAE and AEs were reported in all in one table.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.